CLINICAL TRIAL: NCT03305523
Title: The Safety of Thermocautery Usage for Male Children's Circumcisions
Acronym: MC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocatepe University (Other)
Responsible Party: Principal Investigator, Ahmet Ali Tuncer, Asst Prof Dr, Kocatepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2011-KAEK-2 2017/2:52
Record Dates: First submitted 2017-10-04; First posted 2017-10-10 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Circumcision, Male
Keywords: circumcision; Thermocautery; Complication

STUDY DESIGN:
Intervention Model Description: Short and long-term complications of male circumcisions using thermocautery was examined during 2 years period.
  Complications were classified as perioperative (bleeding during the circumcision or under observation at the hospital after circumcision that required knotting or cauterization, scrotum or penile injury), early postoperative (first 10 days after being discharged) and long-term (late postoperative = after 10 days) (skin-mucosal bridge, delayed wound healing, secondary phimosis, meatitis).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thermocautery (Experimental): Circumcision with thermocautery technique was applied all participants
  Interventions: Device: Thermocautery

INTERVENTIONS:
Device: Thermocautery — In the thermocautery method, a digital thermocautery device (Thermo-Med TM 802-B, Thermo Medical, Adana, Turkey) with 6 different temperature settings was used. Circumcision was performed in the same way as the surgical circumcision. Only cutting and bleeding intervention was done by using a thermocautery device. Cutting was performed by making the appropriate heat adjustment according to the age of the child and the thickness of the glans. Hemorrhage control was performed with a thermocautery device and then the skin-mucosa integrity was ensured by using a 5/0 absorbable suture
  Other Names: Study group

SUMMARY:
Since circumcision is a significant workload for surgeons working at the rural state hospitals in Turkey, the use of circumcision techniques that are easy to implement and have low complications is becoming widespread. This research will examine short and long-term complications of male circumcisions using thermocautery technique in light of current literature.

DETAILED DESCRIPTION:
Patients who were circumcised between May 2014 and May 2016 at the Pediatric Surgery and Urology Clinics at Yuksekova State Hospital were retrospectively analyzed through the hospital registry system. Patients who underwent circumcision with thermocautery technique were examined in terms of age, duration of circumcision and complication rates. Complications were classified as perioperative (bleeding during the circumcision or under observation at the hospital after circumcision that required knotting or cauterization, scrotum or penile injury), early postoperative (first 10 days after being discharged) and long-term (late postoperative = after 10 days) (skin-mucosal bridge, delayed wound healing, secondary phimosis, meatitis).

Patients were discharged after being kept under observation for 1 hour after circumcision. Patients were suggested to apply routine warm sitting bath, daily dressing and the patients with phimosis opening were suggested to apply epithelizing cream. On the 10th postoperative day, all patients were called for control. Patients who developed complications were included in long-term follow-up. Complications were treated.

Statistical analysis: The data obtained from the study were transferred to a computer environment and evaluated with the help of Statistical Package for Social Sciences Version 19.0. Chi-square test was used to evaluate categorical data and Mann-Whitney U test was used to evaluate quantitative variables. P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

Patients who circumcised by Thermocautery device Patients without additional disease between 2 weeks and 18 years included in the study Male gender

Exclusion Criteria:

* Other circumcision Techniques (Conventional surgical, Alis clamp, Tara, Mogen clamp...)
* Patients older than 18 years
* The presence of additional diseases ( such as hematologic disease, diabetes...)
* Patient with hypospadias

Ages: 2 Weeks to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1780 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2014-05-01 (Actual); Study Completion 2016-05-01 (Actual)

PRIMARY OUTCOMES:
Complication rate | perioperative (during circumcision) - 6 months after circumcision
  On the 10th postoperative day, all patients were called for control. Patients who developed complications were included in long-term follow-up. Complications were classified as perioperative (bleeding during the circumcision or under observation at the hospital after circumcision that required knotting or cauterization, scrotum or penile injury), early postoperative (first 10 days after being discharged) and long-term complications (10 days- 2 years).

SECONDARY OUTCOMES:
Surgical processing time | 4-15 minutes
  Surgical processing times were analyzed retrospectively by using the hospital registry system

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Ali Tuncer, Asst Prof Dr, Principal Investigator — Afyon Kocatepe University

IPD SHARING:
Plan to Share IPD: Undecided